CLINICAL TRIAL: NCT01122810
Title: Head to Head Comparison of Multidetector Coronary Tomography and Conventional Coronary Angiogram in the Setting of Systematic Screening of Coronary Vasculopathy After Orthotopic Heart Transplantation.
Brief Title: Scanner and Transplant Heart Patients Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: French Federation of Cardiology (Other)
Responsible Party: Anissa Bouzamondo, French Society of Cardiology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-07
Record Dates: First submitted 2010-03-02; First posted 2010-05-13 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Heart Transplant Patients
Keywords: Diagnostic accuracy of coronary angiography; Transplant heart patients; X-Ray and contrast agent exposure; Coronary stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Coronary scanner — The ECG-gated contrast-enhanced multidetector computed tomography coronary angiography will be performed with a 64 or 256-row CT Philips, Brilliance. The contrast medium mean quantity used is 80-100 ml. The CT scan parameters, adapted to the patient's weight, include 120 kV, 800mA, 0.625 mm slice thickness, 0.42-s rotation time and 0.2 pitch. To determine X-Ray exposure, Dose Length Product (Gycm) will be measured. Reconstruction will be performed at 40 and 75 % of the cycle using ECG gating. A semi quantitative analyse of coronary narrowing will be performed blindly to coronary angiogram results by two experienced radiologists. The CT quality will be determined using a quality scale from 1 to 5. A Calcification score will also be determined. A segment analyse will be performed according to AHA classification. Only more than 1.5 mm diameter vessel segments will be analysed.
  Other Names: 64 ou 256 row coronary computed tomography

SUMMARY:
Coronary vasculopathy remains the leading cause of decreased survival after the first year post-transplantation. It is mainly asymptomatic because of the denervation of the heart transplant. Currently, annual invasive coronary angiogram is performed to ensure the lack of coronary narrowing. But invasive coronary angiography caries risks of serious adverse events and some concern rise from its repetition in that population. Recent advance in coronary multidetector computed tomography (CT) may allow non invasive visualization of the coronary tree. But, it remains unknown if the encouraging data observed in native coronary artery analysis can be extrapolated to transplant heart recipients. Indeed, only very small sample size studies (20 patients) have been conducted in this particular setting. Thus, the investigators decide to assess the diagnostic accuracy of the 64-row CT and 256-row CT compared to the gold standard coronary angiogram in a larger sample size study. The practice aim of this study is to determine if the conventional invasive coronarography can be switched by the 64-row CT or the 256-row CT to assess coronary anatomy especially for the patient without any coronary artery disease (CAD) or those with CAD not suitable for percutaneous coronary intervention.

DETAILED DESCRIPTION:
Background:

Heart transplantation is a major advance in the care of patient with terminal heart failure. But, despite the spectacular prognosis improvement obtained with this treatment, coronary vasculopathy remains the leading cause of decreased survival after the first year post-transplantation (8% of death at 1 year, 42% at 5 years). This coronary artery disease (CAD) has a particular feature involving immunological and inflammatory process, also favoured by classical risk factors in the context of immunosuppression, with rapid and diffuse involvement. Because of the denervation of the transplant heart, it remains mainly asymptomatic and let non invasive stress tests with poor accuracy for CAD screening. It explains the current use of systematic coronary angiogram to transplant heart recipient's survey.

But coronary angiogram remains an invasive technique and exposed to potential serious adverse events.

The recent advance in coronary multidetector computed tomography (CT) may allow non invasive visualization of the coronary tree. Indeed, 64-row CT has already showed its accuracy for the screening of CAD in symptomatic patient in sinus rhythm. However, they are very few studies in the setting of heart transplantation with small sample size and mainly using 16-row CT. Only two small sample size studies (20 patients each) have been conducted using 64-row CT in the setting of heart transplant recipients. None of them compared X-Ray and contrast iodine exposure.

Aim :

Our primary aim is to compare the diagnostic accuracy value of the 64-row CT and 256-row CT to the gold standard (conventional coronary angiogram) in the setting of CAD screening in a large population of heart transplant recipients (= 110 pts). We make the assumption that the sensitivity of CT is enough to allow switching the coronary angiogram by CT for the screening of asymptomatic CAD in heart transplant recipients without CAD or with CAD not suitable for revascularization.

We plan also to compare X-Ray and contrast agent exposure.

Methods :

All the transplant heart patients systematically followed in the cardiovascular and thoracic surgery service will be prospectively included. All the patients will sign the informed consent, then CT will be performed 24 H before the coronary angiogram.

multidetector coronary computed tomography : The Electrocardiogram (ECG)-gated contrast-enhanced multidetector computed tomography coronary angiography will be performed with a 64 or 256-row CT Philips, Brilliance. The contrast medium (Iomeron*, ioméprol, Bracco-Altana Pharma GmbH) mean quantity used is 80-100 ml. The CT scan parameters, adapted to the patient's weight, include 120 kV, 800mA, 0.625 mm slice thickness, 0.42-s rotation time and 0.2 pitch. To determine X-Ray exposure, Dose Length Product (Gycm) will be measured.

After the scan, the reconstruction will be performed at 40 and 75 % of the cycle using ECG gating. Additional reconstructions at different phase can be performed in case of coronary calcification or motion artefacts.

A semi quantitative analyse (N=normal, I=intermediate, S=stenosis) of coronary narrowing will be performed blindly to coronary angiogram results by two experienced radiologists. The CT quality will be determined using a quality scale (scale from 1 to 5).

A Calcification score will also be determined. A segment analyse will be performed according to AHA classification (17 segments model). Only more than 1.5 mm diameter vessel segments will be analysed.

Coronary angiogram :

According to good practice, patients will receive 0.9 % saline serum intravenously at a dose of 1000 ml per 12 H before and 1000 ml per 12 H after contrast medium injection.

Coronary angiogram will be performed according to standard protocol, using radial access with 4 or 5 French sheath under continuous invasive survey of blood pressure and ECG monitoring. The contrast medium quantity used (Hexabrix*, sodium and méglumine ioxaglate, Guerbet) as the X-Ray dose era product (Gy.cm²) will be measured.

Quantitative coronary analysis will be performed by two experienced interventional cardiologists blind to the CT results. Significant stenosis is defined by a > 50% vessel narrowing.

Serum creatinine will be controlled the day before, the day after and 72 H after the coronary angiogram.

Statistical analysis :

Comparison of the two techniques will be done by segments, by artery and by patients with determination of the sensitivity, specificity, positive and negative predictive value of CT for the screening of significant coronary stenosis (> 50%). Statistical analysis will be made with Statview 5.0.

Ethical comity :

All the patient receive and sign an informed consent. The ethical comity (CPP Ile-de-France VI) approves the protocol and the French Society of Cardiology supported the study.

Expected Calendar :

We plan to perform the CT during systematic annual hospitalisation for invasive coronary angiogram. In the cardiovascular department, approximately 8 patients benefit from coronary angiogram per week. Thus we plan to include 110 patients within 30 months, taking in account the exclusion criteria and the availability of both techniques.

ELIGIBILITY:
Inclusion Criteria:

* Transplant heart patients
* Years > 18
* Informed Content

Exclusion Criteria:

* < 18 years old
* Renal failure (Creatinine > 150 µmol/l)
* Patient in complete arrhythmia due to auricular fibrillation
* Patient with a Cardiac Basic frequency > 100 / min
* Iodine Allergy
* Patient hospitalized except the frame of the annual systematic monitoring
* Pregnancy
* People unable to sign the informed content such as major under supervision
* Patients non affiliated to the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
sensitivity of CT : Frequency of stenosis diagnosed by CT in comparison with frequency of stenosis diagnosed by coronarography | Day 1

SECONDARY OUTCOMES:
specificity, positive predictive value, negative predictive value of CT | Day 1
X-Ray and contrast agent exposure | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Barthelemy, MD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France